CLINICAL TRIAL: NCT04382729
Title: Effects of Neuromuscular Electrical Stimulation Therapy on Physical Function in Patients With COVID-19 Associated Pneumonia: Study Protocol of a Randomized Controlled Trial
Brief Title: Neuromuscular Electrical Stimulation in Patients With COVID19 Associated Pneumonia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Turin, Italy (Other)
Collaborators: San Luigi Gonzaga Hospital (Other)
Responsible Party: Principal Investigator, Marco Alessandro Minetto, Associated Professor, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ESC270320
Record Dates: First submitted 2020-05-08; First posted 2020-05-11 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: COVID-19 Pneumonia
Keywords: COVID-19; Fatigue; Muscle Thickness; Neuromuscular Electrical Stimulation; Post-Intensive Care Syndrome; Quadriceps Muscle; Short Physical Performance Battery
MeSH Terms: conditions — COVID-19; Fatigue; postintensive care syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NMES Group (Experimental)
  Interventions: Other: Neuromuscular Electrical Stimulation
- Control Group (Active Comparator)
  Interventions: Other: Physical Therapy Exercise

INTERVENTIONS:
Other: Neuromuscular Electrical Stimulation — The intervention group, in addition to the daily routine physical therapy, receives NMES for 15 days (5 days per week for 3 weeks). NMES is applied bilaterally using an electrical stimulator with pairs of electrodes placed transversally on the quadriceps muscles and on the gastrocnemius muscles. The stimulation protocol consists in the application of symmetrical biphasic rectangular pulses with a frequency of 30 Hz (pulse duration: 400 µs). Stimulation intensity is adjusted daily by the physical therapist to elicit a visible twitch in each muscle. The total duration of the NMES session is 30 min for the first week and 45 min for the second and third week. Stimulation (on) time is 5 s and relaxation (off) time is 15 s, thus eliciting a total of 90 evoked contractions per day during the first week and 135 contractions per day during the second and third week.
  Arms: NMES Group
Other: Physical Therapy Exercise — The control group is subjected to a protocol of physical therapy exercises, applied once a day for 30 minutes (5 days per week for 3 weeks) by the staff physical therapists. It starts with global passive range of motion exercises, followed by active and resistive exercises (including controlled breathing exercises and respiratory muscle training), transfer to the edge of the bed or to a chair, standing and walking.
  Arms: Control Group

SUMMARY:
Neuromuscular electrical stimulation (NMES) has been considered as a promising approach for the early rehabilitation of patients in and/or after the intensive care unit (ICU). Aim of this study is to evaluate the NMES effect on physical function of COVID-19 patients.

DETAILED DESCRIPTION:
This prospective, randomized, controlled, parallel-group, single-blind trial will include 80 patients who had undergone mechanical or non-invasive ventilation following pneumonia-induced respiratory failure. Patients are randomized to a control group (routine physical therapy for 3 weeks) or a NMES group (routine physical therapy plus NMES of quadriceps and gastrocnemius muscles for 3 weeks). The primary outcome is physical performance assessed through the Short Physical Performance Battery (SPPB). Secondary outcomes include independence level, perceived fatigue, muscle strength, rectus femoris thickness, and walking performance. The SPBB and walking performance will be assessed once (after the 3-week intervention period), while all other outcomes will be assessed twice (before and after the intervention).

NMES is a simple and non-invasive technique for muscle strengthening that is usually well tolerated, does not produce adverse effects, requires no or little cooperation from patients and is quite inexpensive. Therefore, proving the effectiveness of NMES therapy for physical and muscle function in COVID-19 patients could support its systematic incorporation in post-ICU rehabilitation protocols of patients presenting with post-intensive care syndrome.

ELIGIBILITY:
Inclusion Criteria:

* age above 18 years
* respiratory (PaO2/FiO2 ratio > 180 mmHg) and hemodynamic stability for at least two days after withdrawal of mechanical ventilation and neuromuscular blocking agents

Exclusion Criteria:

* pregnancy
* known or suspected malignancy in the lower limbs
* body mass index equal or greater than 35 kg/m2
* conditions preventing NMES treatment (e.g., deep vein thrombosis, skin lesions, rhabdomyolysis)
* conditions preventing the outcome assessment (e.g., amputation or inability to transfer independently from bed to chair before hospital admission)
* presence of an implanted cardiac pacemaker or defibrillator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-04-17 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Short Physical Performance Battery (SPPB) Score | 1 week after the intervention
  The SPPB score is a composite measure assessing standing balance (ability to stand for up to 10 seconds with feet positioned in three ways: together side-by-side, semi-tandem and tandem), walking speed (time to complete a 4-m walk), and sit-to- stand performance (time to rise from a chair five times). Each task is scored out of 4 points, with the scores from the three tests summed up to give a total, with a maximum of 12 points and a minimum of 0.

SECONDARY OUTCOMES:
Functional Independence Measure (FIM) Scale Score | Before and 1 week after the intervention
  The FIM is an 18-item, clinician-reported scale that assesses function in six areas including self-care, continence, mobility, transfers, communication, and cognition. Each of the 18 items is graded on a scale of 1-7 based on level of independence in that item (1 = total assistance required, 7 = complete independence)
Fatigue Severity Scale Score | Before and 1 week after the intervention
  The Fatigue Severity Scale is a 9-item scale which measures the severity of fatigue and its effect on a person's activities and lifestyle
Muscle Strength | Before and 1 week after the intervention
  Handgrip strength is assessed for both sides using a handheld device. Patients are instructed to perform a maximal voluntary isometric contraction by contracting their muscles as forcefully as possible for 4-5 s. The test is repeated three times for each side and the highest value is retained. Lower limb strength is assessed as the sum of knee extension and plantar flexion strength of both sides. Muscle strength is rated using the Medical Research Council (MRC) scale that ranges from 0 (no muscle contraction) to 5 (normal resistance), for a maximum score of 20 points.
Two Step Test Length | 1 week after the intervention
  Subjects are required to step out with the dominant leg maximally, then to step out with the other leg maximally, and then to draw and match the first leg to the second leg while maintaining body stability with either supporting leg. The distance between the start line and the tiptoe of the second step foot is measured as the double step length (sum of the first and second steps).
Six Minutes Walking Test Distance | 1 week after the intervention
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
Muscle Thickness | Before and 1 week after the intervention
  Ultrasound-derived muscle thickness is measured as the distance between the superficial and deep aponeuroses of the rectus femoris muscle (that is measured half-way along the line from the anterior-superior iliac spine to the superior border of the patella). Three consecutive static scans of the rectus femoris of both thighs are acquired in the transverse plane and the mean of six measurements (three measurements per side) is considered.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Alessandro Minetto, MD, PhD, Principal Investigator — University of Turin, Italy
Locations (1):
- San Luigi Gonzaga Hospital, Orbassano, TO, Italy

IPD SHARING:
Plan to Share IPD: Yes